CLINICAL TRIAL: NCT02551627
Title: Impact of a Multiple Micronutrient (MMN) Beverage Powder on Vaccine Response in School Children (7-10yrs; Inclusive) in Bangladesh: a Randomised, Double Blind Controlled Trial
Brief Title: A Study to Investigate the Impact of a Multiple Micronutrient (MMN) Beverage Powder on Vaccine Response in School Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 204476
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Growth and Development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product (Experimental): MMN fortified beverage powder [27 gram (g)] made up in 150 milliliter (mL) of water, will be administered orally as a single serve, twice daily for 18 weeks.
  Interventions: Dietary Supplement: Test Product
- Control (Active Comparator): Isocaloric beverage powder without micronutrient fortification (27 g), made up in 150 mL of water will be administered orally as a single serve, twice daily for 18 weeks.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Test Product — MMN fortified beverage powder.
  Arms: Test Product
Dietary Supplement: Control — Isocaloric beverage powder without micronutrient fortification.
  Arms: Control

SUMMARY:
This will be a double blind, two-arm, parallel-group, stratified for gender, randomised, controlled study in participants aged 7-10 years (yrs). The aim of the study is to test the hypothesis that MMN fortified beverage may help improve immunity outcomes as assessed through vaccine response in 7-10 yrs old school participants.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and willingness to participate in the study as demonstrated by participants' parents and/or Legally acceptable representatives (LARs) voluntary written informed consent, participants' written assent
* Participants aged between 7-10 yrs, inclusive
* Good general and mental health
* Participants with Z-scores of BMI for age of ≥-3 to ≤+1

Exclusion Criteria:

* Children in Care (CiC)
* Known or suspected intolerance or hypersensitivity to the study material or any of their stated ingredients or any known food allergies like peanut allergy, gluten allergy or lactose intolerance
* Participant who has already been administered cholera vaccine in any form prior to this study and any known contra-indication to oral cholera vaccine
* Participant who consumed any antibiotics during the week prior to the first dose of study vaccination until the end of the study
* Severe anemia (Hb < 8 g/dL), recent history (2 months) of serious infections, injuries and/or surgeries
* Participant consuming nutritional supplement and/or health food drinks on regular basis (≥ 3 times a week) in last 3 months
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder
* Participants likely to move out of geographical range of the study within study duration
* Child of an employee of the sponsor or the study site or members of their immediate family, sibling of participant already enrolled in the study
* Previous participation in this study, in another clinical study or receipt of an investigational drug within 30 days of screening visit; participation in any nutritional study or didactic nutritional education in last 6 months of the screening visit

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Vaccine response test | 18 weeks
  Proportion of participants demonstrating vaccine reponse, receiving either test product or control will be determined and compared. Vaccine response will be defined as greater than or equal to 4 fold increase from pre-vaccine visit in vibriocidal antibody response 7 days post second vaccine dose.

SECONDARY OUTCOMES:
Absolute vibriocidal antibody titer | 18 weeks
  Blood will be drawn by qualified study personnel as per visits and antibody levels will be assessed.
Change from baseline in nutrional biochemistry | 18 weeks
  Change in nutritional biochemistry for micronutrients vitamins A, B6, B12, C, D, E, folate and of the trace elements (selenium, zinc, copper, iron), ferritin, serum transferrin receptor (sTfR), C-reactive protein (CRP), alpha 1-acid glycoprotein (AGP) from baseline to end of the intervention will be measured from the drawn blood.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline